CLINICAL TRIAL: NCT01951313
Title: EffectEffects of Egg Consumption on Carotenoid Absorption From Co-consumed, Non-Egg Food
Brief Title: Effects of Egg Consumption on Carotenoid Absorption From Co-consumed, Non-Egg Food
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Professor, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 1308013929
Record Dates: First submitted 2013-09-12; First posted 2013-09-26 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Will Consuming Eggs With a Mixed Vegetable Salad Increase Carotenoid Absorption
Keywords: Meal tolerance test focusing on carotenoids absorption

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Egg consumption (Experimental): No egg 75g of scrambled eggs 150g of scrambled eggs
  Interventions: Other: Egg consumption

INTERVENTIONS:
Other: Egg consumption — Subjects will participate in 3 testing days (randomized, crossover design). Each day, the subject will consume a carefully portioned mix-vegetable salad without eggs (C, control); 75g (about 1½ eggs) scrambled whole egg (LE, low egg), and 150g (about 3 eggs) scrambled whole egg (HE, high egg). Prior to each testing day, subjects will consume a low-carotenoid diet for 7 days to reduce blood carotenoid concentration. In the testing day, blood collected every 60 minutes for 10 hours will be processed to analyze carotenoid and vitamin E concentrations. At the 5-h time point, subjects will be fed a low fat (< 2g) and low carotenoid (< 2000µg) meal as the 2nd meal.

SUMMARY:
The 2010 Dietary Guidelines for Americans emphasizes consumption of 4.5 cups of fruits and vegetables daily but average intake of US adults is only 2.6 cups. This low consumption of fruits and vegetables results in limited availability of certain nutrients found in these foods such as carotenoids. Dietary carotenoids have health beneficial properties and are known to fight against disease. Eggs are known to be a good source of carotenoids and eggs may improve the absorption of carotenoids found in co-consumed fruits and vegetables. Therefore, we are interested to see if consuming eggs with a mixed-vegetable salad will increase carotenoid absorption.

DETAILED DESCRIPTION:
The 2010 Dietary Guidelines for Americans emphasizes consumption of 4.5 cups of fruits and vegetables daily. However, average fruit and vegetable intake of US adults is only 2.6 cups. This low consumption of fruits and vegetables may further result in the limited availability of fat soluble, health-promoting, phytochemicals such as carotenoids from these foods. Dietary carotenoids have beneficial biological properties including antioxidant and anti-inflammatory effects and scientific research supports the protective effects of carotenoids against many degenerative diseases, including cardiovascular diseases, age-related macular degeneration, and some types of cancer. Therefore, either low intake or inefficient bioavailability of carotenoids from fruits and vegetables may reduce their potential effectiveness as disease preventative compounds. The bioavailability of carotenoids from a meal can be affected by several factors, including food matrix, type of food processing or cooking, interactions with other dietary compounds during digestion and absorption, gut status which may affect digestion and absorption processes, and nutritional status. Co-consumption of carotenoid rich foods with dietary lipids may be one of the most effective stimulators of carotenoid absorption among factors that influence their bioaccessibility and bioavailability. Eggs are known to be a highly bioavailable source of carotenoids, presumably due to the presence of lipid and phospholipid in egg yolk. The highly bioavailable nature of carotenoids from eggs suggest that egg derived factors may be leveraged to improve bioavailability of other carotenoids found in co-consumed fruits and vegetables. While promising, very limited data exist on the impact of a co-consumed food source of lipid, such as eggs, to enhance carotenoid absorption. This study is designed to assess the beneficial effects of egg consumption on carotenoids absorption from a complex meal, beyond those found in egg.

ELIGIBILITY:
Inclusion Criteria:

Male 19 to 45y BMI 18.5-29.9kg/m2 generally healthy non-smoker

Exclusion Criteria:

Female deep vein thrombosis intestinal disorders fasting blood glucose >110mg/dL smoking drinking more than 3 alcoholic drinks per day taking lipid-lowering medications or dietary supplements affecting plasma cholesterol concentration.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Carotenoids absorption | 6-8 weeks
  Carotenoids absorption Area under the curve of carotenoids such as lutein, zeaxanthin, α-carotene, α-cryptoxanthin, β-cryptoxanthin, β-carotene, and lycopene and vitamin E in plasma triacylglycerol rich lipoproteins fractions

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph.D, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Kim JE, Ferruzzi MG, Campbell WW. Egg Consumption Increases Vitamin E Absorption from Co-Consumed Raw Mixed Vegetables in Healthy Young Men. J Nutr. 2016 Nov;146(11):2199-2205. doi: 10.3945/jn.116.236307. Epub 2016 Sep 21. PMID 27655756
- [Derived] Kim JE, Gordon SL, Ferruzzi MG, Campbell WW. Effects of egg consumption on carotenoid absorption from co-consumed, raw vegetables. Am J Clin Nutr. 2015 Jul;102(1):75-83. doi: 10.3945/ajcn.115.111062. Epub 2015 May 27. PMID 26016861